CLINICAL TRIAL: NCT02029404
Title: Approach to Continuous Sciatic Nerve Block for Orthopedic Procedures in Day Surgery With Two Different Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Andrea Luigi Ambrosoli, Chief of Day Surgery department Ospedale di Circolo Varese, Ospedale di Circolo - Fondazione Macchi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAA-001
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2014-10

CONDITIONS: Regional Anesthesia Morbidity; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tibial nerve group (Active Comparator): In the TN (tibial nerve ) group probe will be placed in popliteal cave to identify the popliteal artery and laterally the tibial nerve. Identified the tibial nerve we will proceed , previous local anaesthesia, to insert a catheter medially to tibial branch of the sciatic nerve according to in plane approach.
  Interventions: Procedure: Tibial nerve group
- Tibial peroneal nerve group (Active Comparator): In the TPN (tibial -peroneal nerve) group the probe will be placed in popliteal cave to identify the popliteal artery and laterally the tibial nerve. Afterwards, proceeding cranially with the probe according to "in plane" approach, we will identify the confluence of tibial with peroneal branch and in this point, previous local anaesthesia, we will position the catheter within the confluence of peroneal and tibial nerve.
  Interventions: Procedure: Tibial peroneal nerve group

INTERVENTIONS:
Procedure: Tibial nerve group — After the recovery of the sensitivity we will start the continuous infusion of levobupivacaine 0,125% with a portable pump (Mini Rythmic Evolution, Micrel Medical Devices) with a flow basal rate 2 ml/h and a rescue bolus doses of 2 ml (lock out 20 minutes). Before the discharge from the hospital, if the NRS will be > 4, a bolus of 10 ml of Mepivacaine 1% through the catheter could be administered.
  An "information sheet" will be released at the discharge and the medical indication for any "rescue doses" at home.
  The patients will be contacted by phone at POD 1-2 and will allowed to answer to a questionnaire (see endpoint) At POD 3 the patients will come in our ambulatory where we will remove the catheter and they will return the pump
  Arms: Tibial nerve group
Procedure: Tibial peroneal nerve group — After the recovery of the sensitivity we will start the continuous infusion of levobupivacaine 0,125% with a portable pump (Mini Rythmic Evolution ,Micrel Medical Devices )with a flow basal rate 2 ml/h and a rescue bolus doses of 2 ml (lock out 20 minutes). Before the discharge from the hospital, if the NRS will be > 4, a bolus of 10 ml of Mepivacaine 1% through the catheter could be administered.
  An "information sheet" will be released at the discharge and the medical indication for any "rescue doses" at home.
  The patients will be contacted by phone at POD 1-2 and will allowed to answer to a questionnaire (see endpoint) At POD 3 the patients will come in our ambulatory where we will remove the catheter and they will return the pump
  Arms: Tibial peroneal nerve group

SUMMARY:
We will enroll patients submitted to feet elective orthopaedic surgery that require analgesia through continuous peripheral nerve block (CNPB) of the sciatic nerve. All catheters will be placed by anaesthesiologists experienced in ultrasound in prone positioning. The patients will be randomized in two groups with technique of sealed envelopes.

In the tibial -peroneal nerve (TPN) group we will position the catheter within the confluence of peroneal and tibial nerve.

In the tibial nerve (TN) group we will proceed , previous local anaesthesia, to insert a catheter medially to tibial branch of the sciatic nerve according to in plane approach.

We will analyze A: the difference in consumption of local anesthetic in the two different groups B: the difference of "insensate limb" in the post-operative home as described by Ilfeld(inability to perceive the sense of touch throughout the area of distribution of the sciatic nerve) C: rate of foot drop D: numeric rate scale (NRS) for pain assessment, rate of dislodgment of the catheters, patient satisfaction, need for intervention by the anesthesiologist after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates for orthopedic surgery of the lower limb in unilateral day-surgery with surgical incision in the distribution of the sciatic nerve
* Patients according to American Society of Anesthesiologists scale (ASA) I-II
* Age greater than 18 years
* Informed Consent
* Presence of a "caretaker" for the night and the next day.

Exclusion Criteria:

* Contraindications to regional anesthesia
* Patients ASA III-IV
* Patients receiving therapy for chronic pain
* Patients with: renal failure, coagulopathy, liver failure, peripheral neuropathy
* Refusal by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Compare the difference in consumption of local anesthetic in the two different groups | within the first two days after surgery

SECONDARY OUTCOMES:
Analyze the difference of "insensate limb"in the post-operative home as described by Ilfeld (inability to perceive the sense of touch throughout the area of distribution of the sciatic nerve) | within the first two days after surgery

OTHER OUTCOMES:
analyze the rate of foot drop in these two different groups | within the first two days after surgery
analyze the NRS in these two different groups | within in the first two days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Luca Guzzetti, MD, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- Department of Day Surgery Ospedale di Circolo Varese, Varese, VA, Italy